CLINICAL TRIAL: NCT07165548
Title: Evaluation of the Effect of Supplementation With Satiating Compounds Integrated Into a Hypocaloric Diet on Weight and Cardiometabolic and Osteoarticular Health in Overweight/Obese Subjects
Brief Title: Impact of Satiating Compounds and Hypocaloric Diet on Weight, Cardiometabolic and Osteoarticular Health in Obesity
Acronym: COGLUBOCO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COGLUBOCO (2025.116)
Record Dates: First submitted 2025-08-28; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Obesity; Overweight
Keywords: Nutritional intervention; Dietary supplement; Protein bar; Fiber bar; Hypocaloric Diet; Obesity; Weight loss; Satiety; Cardiometabolic health; Osteoarticular health; Quality of life
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

STUDY DESIGN:
Intervention Model Description: 4 parallel groups, 12-week, randomized nutritional intervention
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Experimental group 1 (Experimental): Bars containing satiating compounds: formulation 1
  Interventions: Dietary Supplement: Experimental Bar (Formulation 1) + Hypocaloric diet (10% energy restriction)
- Experimental group 2 (Experimental): Bars containing satiating compounds: formulation 2
  Interventions: Dietary Supplement: Experimental Bar (Formulation 2) + Hypocaloric diet (10% energy restriction)
- Experimental group 3 (Experimental): Bars containing satiating compounds: formulation 3
  Interventions: Dietary Supplement: Experimental Bar (Formulation 3) + Hypocaloric diet (10% energy restriction)
- Placebo group (Placebo Comparator): Placebo bars
  Interventions: Dietary Supplement: Placebo Bar + Hypocaloric diet (10% energy restriction)

INTERVENTIONS:
Dietary Supplement: Experimental Bar (Formulation 1) + Hypocaloric diet (10% energy restriction) — Participants will consume three satiating compound-enriched bars (formulation 1) daily, 30 minutes before breakfast, lunch, and dinner, as part of a 10% energy-restricted hypocaloric diet for 12 weeks.
  Arms: Experimental group 1
Dietary Supplement: Experimental Bar (Formulation 2) + Hypocaloric diet (10% energy restriction) — Participants will consume three satiating compound-enriched bars (formulation 2) daily, 30 minutes before breakfast, lunch, and dinner, as part of a 10% energy-restricted hypocaloric diet for 12 weeks.
  Arms: Experimental group 2
Dietary Supplement: Experimental Bar (Formulation 3) + Hypocaloric diet (10% energy restriction) — Participants will consume three satiating compound-enriched bars (formulation 3) daily, 30 minutes before breakfast, lunch, and dinner, as part of a 10% energy-restricted hypocaloric diet for 12 weeks.
  Arms: Experimental group 3
Dietary Supplement: Placebo Bar + Hypocaloric diet (10% energy restriction) — Participants will consume three placebo bars daily, 30 minutes before breakfast, lunch, and dinner, as part of a 10% energy-restricted hypocaloric diet for 12 weeks.
  Arms: Placebo group

SUMMARY:
The main objective of this intervention study is to evaluate the effect of satiating protein and/or fiber bar consumption on weight loss and other osteoarticular and cardiometabolic parameters related to excess weight in subjects with overweight or obesity.

To achieve this objective, volunteers will be instructed to consume three bars per day as part of a hypocaloric diet, in accordance with healthy nutritional guidelines, over a 12-week period.

The main questions to answer are:

* Does the regular consumption of these protein and/or fiber bars help to lose weight?
* Does the regular consumption of these protein and/or fiber bars help to improve the osteoarticular health?
* Does the regular consumption of these protein and/or fiber bars help to improve the cardiometabolic health?

The specific objectives are focused on evaluating the effects of the intervention on the following parameters:

* Weight and body composition.
* Knee joint range of motion.
* Blood biomarkers related to collagen degradation and synthesis, associated with osteoarticular health.
* Glycemic and lipid profiles, blood pressure, and biomarkers of kidney, liver, cardiovascular, and inflammatory health.
* Changes in joint discomfort (improvement or worsening).
* Adherence to the assigned intervention, including both dietary compliance and intake of the study-provided supplement.
* Satiety-related variables assessed using a visual analog scale (VAS).
* Urinary hydroxyproline and stool samples for metagenomic analysis.
* Gastrointestinal health, mental health, quality of life, and physical activity level assessed through validated questionnaires.

Target sample size is 144 subjects and participants will be allocated in four different groups:

* Group 1 (n=36): hypocaloric diet + protein and fiber supplement.
* Group 2 (n=36): hypocaloric diet + protein and fiber supplement.
* Group 3 (n=36): hypocaloric diet + fiber supplement.
* Group 4 "Placebo group" (n=36): hypocaloric diet + placebo supplement. Participants will attend the nutritional intervention unit at weeks 1, 8, and 12. A follow-up phone call will be conducted at week 4.

DETAILED DESCRIPTION:
Volunteers expressing interest in the study will undergo an initial eligibility assessment, either via telephone interview or by completing an online screening form (Google Form), to verify compliance with the primary inclusion criteria. Candidates meeting these criteria will be invited to attend an information and screening visit, during which the study procedures will be explained in detail and any questions addressed. Individuals who agree to participate will provide written informed consent and will be randomly allocated to one of the four intervention groups. All necessary study materials will be provided at this stage.

Participants will attend three scheduled clinical investigation visits: baseline (day 0), mid-intervention (week 8), and post-intervention (week 12). At each visit, anthropometric and body composition measurements will be performed, and blood pressure will be recorded. Biological samples, including blood, urine, and stool, will be collected. In addition, data regarding dietary intake, physical activity levels, sleep patterns, and gastrointestinal symptoms will be obtained through validated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers of both sexes between the ages of 18 and 65 years old.
* Volunteers with grade II overweight or obesity (BMI: 27.0-39.9 kg/m2).
* Physical examination and vital signs are normal or clinically irrelevant to the study.
* Volunteers receiving pharmacological treatment may be included if the dosage has remained stable for at least three months prior to study initiation.
* Individuals undergoing treatment for diabetes will be excluded.
* Participants must be capable of understanding the study requirements, willing to provide written informed consent, and able to comply with all study procedures and timelines.
* Body weight must have remained stable (±5%) during the three months preceding study initiation.

Exclusion Criteria:

* Presence of significant functional or structural abnormalities of the digestive system, including but not limited to congenital malformations, angiodysplasia, active peptic ulcer disease, chronic inflammatory or malabsorption disorders, hiatal hernia, or chronic gastroesophageal reflux.
* High alcohol consumption, defined as >14 units per week for women and >20 units per week for men.
* Pregnancy or lactation at the time of screening.
* History of surgical procedures resulting in permanent alterations of the digestive system (e.g., gastroduodenostomy) or joint replacement surgery (hip or knee).
* Diagnosis of arthritis.
* History of any liver disease, with the exception of non-alcoholic fatty liver disease.
* Diagnosis of any type of cancer, current cancer treatment, or history of cancer treatment within the past five years.
* Known allergy or hypersensitivity to any component of the investigational product or to any food that could interfere with study participation and follow-up.
* Presence of cognitive and/or psychological impairment that could affect study compliance.
* Anticipated poor adherence or, in the opinion of the investigator, inability to comply with study procedures.
* Engagement in night-shift work.
* Current use of dietary supplements that may interfere with study outcomes (e.g., nutraceuticals containing compounds with potential weight loss effects).
* Ongoing treatment for weight loss or diabetes.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Body weight | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Weight of participants will be measured by bioimpedance an densitometry and reported in kg

SECONDARY OUTCOMES:
Height | Clinical Investigation Day 1
  Height of participants will be measured by stadiometer and reported in cm.
Body mass index | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Body mass index will be calculated as follows: weight (kilograms)/ height (m)2
Waist circumference | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Waist circumference of participants in fasting condition will be analyzed by measuring tape and reported in centimeters.
Hip circumference | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Hip circumference of participants in fasting condition will be analyzed by measuring tape and reported in centimeters.
Neck circumference | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Neck circumference of participants in fasting condition will be analyzed by measuring tape and reported in centimeters.
Body fat mass | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Body fat of participants will be analyzed by bioimpedance and densitometry and reported in percentage and kilograms.
Body lean mass | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Body lean mass of participants will be analyzed by bioimpedance and densitometry and reported in kilograms.
Body muscle mass | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Body muscle mass of participants will be analyzed by bioimpedance and densitometry and reported in kilograms.
Fat free mass | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3.
  Fat free mass of participants will be analyzed by densitometry and reported in kilograms.
Visceral fat | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Visceral fat of participants will be measured by bioimpedance an densitometry and reported in g.
Body water mass | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Body water mass of participants will be analyzed by bioimpedance and densitometry and reported in kilograms and percentage.
Body bone mass | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Body bone mass Body bone mass of participants will be analyzed by bioimpedance and densitometry and reported in kilograms.
Systolic blood pressure | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Systolic blood pressure of participants in fasting condition will be analyzed by electronic tensiometer and reported in mmHg
Diastolic blood pressure | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Diastolic blood pressure of participants in fasting condition will be analyzed by electronic tensiometer and reported in mmHg
Heart rate | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Heart rate of participants in fasting condition will be analyzed by electronic tensiometer and reported in pulses/min.
Total bone mineral density | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Total bone mineral density of participants will be analyzed by densitometry and reported in g/cm2.
Bone mineral density L1-L4 | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3.
  Bone mineral density L1-L4 of participants will be analyzed by densitometry and reported in g/cm2.
Total bone mineral density femur | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3.
  Total bone mineral density femur of participants will be analyzed by densitometry and reported in g/cm2.
Bone mineral density femur neck | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3.
  Bone mineral density femur neck of participants will be analyzed by densitometry and reported in g/cm2.
Knee articular range | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3.
  Knee articular range of participants will be measured using a goniometer and performing the chair test.
Grip strength | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3.
  Grip strength of participants will be measured using a manual dynamometer and reported in kg.
Level of hunger | Clinical Investigation Day 1, Clinical Investigation Day 2
  Hunger of participants will be analyzed by Hunger-Satiety Visual Analogue Scale (VAS). The minimum value of the scale is 0 mm and the maximum value is 100 mm. A reduction in hunger scale means better outcome.
Level of fullness | Clinical Investigation Day 1, Clinical Investigation Day 2
  Fullness of participants will be analyzed by Hunger-Satiety Visual Analogue Scale. The minimum value of the scale is 0 mm and the maximum value 100 mm. An incrementation in fullness scale means better outcome.
Level of satisfaction | Clinical Investigation Day 1, Clinical Investigation Day 2
  Satisfaction sensation of participants will be analyzed by Hunger-Satiety Visual Analogue Scale. The minimum value of the scale is 0 mm and the maximum value 100 mm. An incrementation in satisfaction scale means better outcome.
Want to eat something else | Clinical Investigation Day 1, Clinical Investigation Day 2
  Want to eat something else sensation of participants will be analyzed by Hunger-Satiety Visual Analogue Scale. The minimum value of the scale is 0 mm and the maximum value 100 mm. A reduction in want to eat something else scale means better outcome.
Thirst | Clinical Investigation Day 1, Clinical Investigation Day 2
  Thirst sensation of participants will be analyzed by Hunger-Satiety Visual Analogue Scale. The minimum value of the scale is 0 mm and the maximum value 100 mm.
Life quality | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Life quality of participants will be evaluated by SF-36 questionnaire (36-Item Short Form Survey).
Depression | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Depression will be evaluated using the Beck Depression Inventory-II (BDI-II), a 21-item self-report questionnaire. Total scores range from 0 to 63, with higher scores indicating greater severity of depressive symptoms.
Anxiety | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Anxiety will be evaluated using the State-Trait Anxiety Inventory (STAI), a 40-item self-report questionnaire that includes two subscales: State Anxiety (20 items) and Trait Anxiety (20 items). Each subscale yields scores ranging from 20 to 80, with higher scores indicating greater levels of anxiety.
Osteoarticular health | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Osteoarticular health of participants will be measured using the Western Ontario and McMaster Universities Arthritis Index (WOMAC), a 24-item self-report questionnaire that assesses pain (range 0-20), stiffness (range 0-8), and physical function (range 0-68). The total score ranges from 0 to 96, with higher scores indicating worse osteoarticular symptoms and functional impairment.
Physical activity | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Physical activity will be evaluated using the Physical Activity Questionnaire of the Seguimiento Universidad de Navarra (SUN) cohort, which estimates total physical activity expressed in Metabolic Equivalent of Task hours per week (MET-h/week). Higher values indicate greater levels of physical activity. Participants can also be classified into categories of low, moderate, or high physical activity according to standardized SUN cohort scoring procedures.
Gastrointestinal symptoms | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Gastrointestinal symptoms will be registrated through Gastrointestinal Symptoms Rating Scale questionnaire, which is a questionnaire of 15 items. The questionnaire has a seven-point graded likert-type scale, where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms.
Glucose concentration | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Blood glucose levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in mg/dL.
Insulin concentration | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Blood insulin concentration will be analyzed after an overnight fast by ELISA kit and reported in μUI/ml.
HOMA index (Homeostatic Model Assessment Index) | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  HOMA index will be calculated as follows: HOMA-IR (Homeostatic Model Assessment for Insulin Resistance)= [fasting glucose (mmol/L) x fasting insulin (μU/ml)] / 22.5.
Total cholesterol | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Blood total cholesterol levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in mg/dL
HDL cholesterol | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Blood HDL cholesterol levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in mg/dL
LDL cholesterol | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  LDL cholesterol levels of participants in fasting condition will be analyzed by Friedewald formula and reported in mg/dL.
Triglyceride concentration | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Triglyceride levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in mg/dL.
Alanine aminotransferase | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Alanine aminotransferase levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in UI/L.
Aspartate aminotransferase | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Aspartate aminotransferase levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in UI/L.
Gamma-glutamyl transferase | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Gamma-glutamyl transferase levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in UI/L.
Fatty liver Index (FLI) | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Fatty liver Index will be calculated as follows FLI = (e 0.953 × ln (triglycerides) + 0.139 × BMI + 0.718 × ln (ggt) + 0.053 × waist circumference - 15.745)/ (1 + e 0.953 × ln (triglycerides) + 0.139 × BMI + 0.718 × ln (ggt) + 0.053 × waist circumference - 15.745) × 100
Fructosamine concentration | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Blood fructosamine concentration will be analyzed after an overnight fast by ELISA kit and reported in µg/L.
Leptine | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Blood leptine concentration will be analyzed after an overnight fast by ELISA kit and reported in ng/ml
Adiponectin | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Blood adiponectin concentration will be analyzed after an overnight fast by ELISA kit and reported in ng/ml.
Homocysteine | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Blood homocysteine concentration will be analyzed after an overnight fast by biochemical autoanalyzer and reported in μmol/L.
MCP1 (Monocyte Chemoattractant Protein-1) | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Blood MCP1 concentration will be analyzed after an overnight fast by ELISA kit and reported in pg/ml.
TNF-alpha (tumor necrosis factor alpha) | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  TNF-alpha will be analyzed after an overnight fast by ELISA kit and reported in pg/ml.
Interleukin 6 (IL6) | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Blood IL6 concentration will be analyzed after an overnight fast by ELISA kit and reported in pg/ml.
C Reactive protein (CRP) | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Blood CRP concentration will be analyzed after an overnight fast by ELISA kit and reported in mg/L
Blood glycated hemoglobin | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Fasting blood glycated hemoglobin will be reported in percentage.
Plasma CTX-II levels (C-terminal telopeptide of type II collagen) | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Plasma CTX-II levels will be analyzed after an overnight fast by ELISA kit and reported in ng/ml
Plasma C2C levels (Cartilage Collagen Neoepitope) | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3.
  Plasma C2C levels will be analyzed after an overnight fast by ELISA kit and reported in ng/ml.
Plasma CP2 levels (type II procollagen carboxy-propeptide) | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3.
  Plasma CP2 levels will be analyzed after an overnight fast by ELISA kit and reported in ng/ml.
Albumin concentration | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Albumin levels of participants in fasting condition will be analyzed in urine by biochemical autoanalyzer and reported in mg/dl.
Creatinine concentration | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Creatinine levels of participants in fasting condition will be analyzed in urine by biochemical autoanalyzer and reported in mg/dl.
Hydroxyproline | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Urine hydroxyproline concentration will be analyzed after an overnight fast by colorimetry technique and reported in mg/ml.
Blood untargeted metabolomics | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Untargeted metabolites will be expressed and analyzed in plasma and serum according to their intensity measured in arbitrary units (UA), which carries a direct relation with its concentration.
Urine untargeted metabolomics | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Untargeted metabolomics will be expressed and analyzed in urine according to their intensity measured in arbitrary units (UA), which carries a direct relation with its concentration.
Lipidomic | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Lipidomic will be expressed and analyzed in plasma and serum according to their intensity measured in arbitrary units (UA), which carries a direct relation with its concentration.
Dietary Intake (Energy and Nutrients) | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Dietary intake will be assessed using the Food Frequency Questionnaire (FFQ). Outcomes will include energy intake (kcal/day), macronutrient intake (g/day), and micronutrient intake (mg/day or µg/day).
Mediterranean Diet Adherence | Clinical Investigation Day 1, Clinical Investigation Day 2 and Clinical Investigation Day 3
  Adherence to the Mediterranean dietary pattern will be evaluated using the Mediterranean Diet Adherence Questionnaire, with scores ranging from 0 to 14 points. Higher scores indicate greater adherence to the Mediterranean diet.
Snacking frequency | Clinical Investigation Day 1, Clinical Investigation Day 2, and Clinical Investigation Day 3
  Snacking behavior will be recorded using a daily snacking record. Results will be expressed as number of snacks per day.
Adherence to bars consumption | Clinical Investigation Day 2 and Clinical Investigation Day 3
  Adherence will be assessed using the bars consumption record form.
Acceptance of bars | Clinical Investigation Day 3
  Acceptance will be assessed using the acceptance consumption record form.

CONTACTS AND LOCATIONS:
Overall Officials: María Ángeles Zulet, PhD, Principal Investigator — Center for Nutrition Research; Fermín Milagro, PhD, Study Chair — Center for Nutrition Research; Idoia Ibero, Study Chair — Center for Nutrition Research; María Hernández, Study Chair — Center for Nutrition Research; Miguel López, PhD, Study Chair — Center for Nutrition Research; Verónica Ciaurriz, Study Chair — Center for Nutrition Research; Carlos J González, PhD, Study Chair — Center for Nutrition Research; Salomé Pérez, Study Chair — Center for Nutrition Research; Marián Pueyo, Study Chair — Center for Nutrition Research
Locations (1):
- Center for Nutrition Research, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No